CLINICAL TRIAL: NCT03524638
Title: Visbiome Effect on Colorectal Anastomosis and Local Recurrence
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator decided to withdraw the study.
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Russell Farmer, Principal Investigator, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18-0282
Record Dates: First submitted 2018-05-02; First posted 2018-05-15 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM A (Active Comparator): Colorectal surgery with administration of Visbiome
  Interventions: Other: Visbiome; Procedure: Colorectal Surgery
- ARM B (Active Comparator): Colorectal Surgery alone
  Interventions: Procedure: Colorectal Surgery

INTERVENTIONS:
Other: Visbiome — Colorectal surgery plus administration of Visbiome on post-operative day 2.
  Arms: ARM A
Procedure: Colorectal Surgery — Colorectal surgery alone

SUMMARY:
Determine whether the administration of Visbiome after colorectal surgery has any effect on anastomotic leak and local recurrence

DETAILED DESCRIPTION:
Randomized study of Visbiome after colorectal surgery. Subjects will be randomized 1:1 to either VSL3 or no VSL3.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Diagnosis of biopsy proven rectal cancer (CT/MRI)
* Willing and able to comply with protocol requirements
* Able to tolerate surgery
* Able to comprehend and have signed the Informed Consent
* Absence of metastatic disease
* Clinical performance status of ECOG 0 or 1
* Life expectancy of greater than 3 months
* Planned ileostomy as part of their routine care

Exclusion Criteria:

* Severe or refractory ulcerative colitis defined as Mayo Score of greater than or equal to 10, endoscopic disease activity score 3
* Untreated enteric infection (positive stool test for any of the following: clostridium difficile, salmonella, shigella, yersinia, campylobacter, enteropathogenic E. coli or other enteric infection at the discretion of the Investigator
* Severe immunodeficiency, inherited or required (e.g. HIV, chemotherapy or radiation therapy)
* Patients with the following laboratory abnormalities: absolute neutrophil count <1000/ul, platelets <50 x 10^9/L, hemoglobin <6.5g/dL
* History of anaphylaxis (severe allergic reaction) to food allergens (e.g. tree nuts, shellfish)
* Active intestinal obstruction
* Non-steroidal anti inflammatory medications (NSAIDs) as long-term treatment, defined as for at least 4 days per week each month
* Cholestyramine use
* Any condition in which the Investigator thinks VSL3 administration may pose a health risk (e.g. severely immunocompromised)
* Simultaneous participation in another interventional clinical trial
* Patients who are pregnant, breast feeding or planning pregnancy during study trial period
* Patients with any other signification medical condition that could confound or interfere with evaluation of safety, tolerability or prevention compliance with the study protocol at the discretion of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2019-07-29 (Actual)

PRIMARY OUTCOMES:
Development of Anastomotic Leak | Hospital discharge, 2 and 4 weeks post-treatment. Then every 3 months for 1 year.
  Development of anastomotic leak will be evaluated by sigmoidoscopy
Local Recurrence | Every three months for 1 year post hospital discharge.
  CT scans will be performed every 3 months after hospital discharge to check disease status

IPD SHARING:
Plan to Share IPD: No